CLINICAL TRIAL: NCT03725579
Title: Anesthetic Efficacy of 2% Mepivacaine Versus 4% Articaine for Inferior Alveolar Nerve Blocks in Patients With Symptomatic Irreversible Pulpitis in Mandibular Molars: A Randomized Clinical Trial PART 6
Brief Title: Anesthetic Efficacy of 2% Mepivacaine Versus 4% Articaine
Acronym: Anesthesia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Mahmoud Bedier, Lecturer in Endodontics Département, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CEBD-CU-2014-06-01
Record Dates: First submitted 2018-10-23; First posted 2018-10-31 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: Anesthetic efficacy; Inferior alveolar nerve blocks

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mepivacaine hydrochloride (Experimental): 2% Mepivacaine hydrochloride with 1:100,000 epinephrine anaesthetic solution. Each patient received two inferior alveolar nerve block injections of the tested anesthetic solution by using a side loading aspirating syringe and 27-gauge long needle
  Interventions: Drug: mepivicane hydrochloride; Drug: articane hydrochloride
- articaine hydrochloride (Active Comparator): 4 % Articaine hydrochloride with 1:100,000 epinephrine anaesthetic solution. Each patient received two inferior alveolar nerve block injections of the tested anesthetic solution by using a side loading aspirating syringe and 27-gauge long needle
  Interventions: Drug: mepivicane hydrochloride; Drug: articane hydrochloride

INTERVENTIONS:
Drug: mepivicane hydrochloride — Pain will be assessed during access cavity preparation and instrumentation
  Other Names: mepivicane
Drug: articane hydrochloride — Pain will be assessed during access cavity preparation and instrumentation
  Other Names: articane

SUMMARY:
The aim of this prospective randomized clinical trial was compare between 2% Mepivacaine and 4% Articaine for inferior alveolar nerve blocks in patients with symptomatic irreversible pulpitis in mandibular molars as regards to their anesthetic efficiency; during access cavity preparation and instrumentation.

DETAILED DESCRIPTION:
Sixty-six patients diagnosed clinically and radiographically with symptomatic irreversible pulpitis in mandibular posterior teeth will received single-visit root canal treatment using ProTaper Universal rotary system for canal preparation, then they will be randomly divided into two groups (n=33) according to the anesthetic solution used, either Group M (3.6 ml Mepivacaine hydrochloride 2% with 1:100000 epinephrine) or Group A (3.4 ml Articaine hydrochloride 4% with 1:100000 epinephrine). The pain will be assessed using numerical rating scale (NRS) during access cavity preparation and instrumentation, then the need for supplemental anesthesia will be also recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in good health (American Society of Anesthesiologists Class II or higher)
2. Patients having symptomatic irreversible pulpitis in one of their mandibular molars.
3. Age range is between 20 and 50 years.
4. Patients who can understand Visual Analogue Scales VAS.
5. Patients able to sign informed consent

Exclusion Criteria:

1. Patients allergic to articaine and/or mepivacaine and/or sulfur
2. Patients having active sites of pathosis in the area of injection.
3. Patients having active pain in more than one molar.
4. Patients who had taken analgesics in the 12 hours preceding the injection.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity: Numerical rating scale (NRS) | Fifteen minutes after injection of the anaesthetic solution
  Pain intensity during access cavity preparation using numerical rating scale (NRS). The scale was numerical to facilitate its use by the participants. The Numerical rating scale is an 10-point scale anchored by two extremes "No pain" and "pain as bad as it could be".
  Pain was categorized into four categorical scores: (1) none [score 0], (2) mild [score from 1-3], (3) moderate [score from 4-6], (4) severe [score from 7-10].

SECONDARY OUTCOMES:
Pain intensity: Numerical rating scale (NRS) | Twenty-five minutes after injection of the anaesthetic solution
  Pain intensity during root canal negotiation and instrumentation using Numerical rating scale is an 10-point scale anchored by two extremes "No pain" and "pain as bad as it could be".
  Pain was categorized into four categorical scores: (1) none [score 0], (2) mild [score from 1-3], (3) moderate [score from 4-6], (4) severe [score from 7-10].
The number of patients who need suplemental anesthesia | Fifteen minutes after injection of the anaesthetic solution
  counting the number of the number of patients who need suplemental anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Bedier, PHD, Study Director — Cairo university, faculty of dentistry
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided